CLINICAL TRIAL: NCT03034603
Title: The Safety and Efficacy Test of Nutri-PEITC Jelly in Head and Neck Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dental Innovation Foundation Under Royal Patronage (Other)
Collaborators: Mahidol University (Other); Srinakharinwirot University (Other); Ministry of Health, Thailand (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: DIF-04
Record Dates: First submitted 2017-01-25; First posted 2017-01-27 (Estimated); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: Head and Neck Neoplasms; Quality of Life; Nutrition Related Cancer
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — phenethyl isothiocyanate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nutri-jelly with PEITC (Experimental): Continuous intake of 200 g Nutri-jelly with 20 mg PEITC per day, five days per week for 3 months.
  Interventions: Dietary Supplement: Nutri-jelly with PEITC
- Nutri-jelly (Placebo Comparator): Continuous intake of 200 g Nutri-jelly per day, five days per week for 3 months.
  Interventions: Dietary Supplement: Nutri-jelly

INTERVENTIONS:
Dietary Supplement: Nutri-jelly with PEITC — Nutri-jelly with PEITC resulted from an addition of tested amount of PEITC, which was shown in animal model to delay cancer growth, into Nutri-jelly.
  Arms: Nutri-jelly with PEITC
Dietary Supplement: Nutri-jelly — Nutri-jelly is an edible nutritious gel for patients with chewing and swallowing difficulties. One milligram of Nutri-jelly contains approximately 1 kcal.
  Arms: Nutri-jelly

SUMMARY:
This triple-blinded randomized placebo control trial aims to investigate the safety and efficacy of Nutri-PEITC jelly, a functional food, in head and neck cancer patients. The primary outcome measure includes adverse events, health-related quality of life, tumor response and progression-free survival. The secondary outcome includes serum p53 and cytochrome C levels and functional status.

DETAILED DESCRIPTION:
Previously, Nutri-jelly, a novel edible nutritious gel for patients with chewing and swallowing difficulties, was shown to be effective in improving the quality of life of head and neck cancer patients. Recently, Nutri-PEITC jelly is recently developed by addition of Phenethyl Isothiocyanate (PEITC), a phytochemical compound with chemopreventive action in animal bearing oral cancer. It intends to be a functional food for cancer survivor. The dose of PEITC in Nutri-jelly was based on safe and effective dose determined in animal studies. Furthermore, Nutri-PEITC jelly was proven safe in healthy volunteers who daily consumes for a consecutive month with no serious adverse events. The purpose of this study is to determine safety and efficacy of Nutri-jelly with PEITC in head and neck cancer patients.

independent variable: continuous Nutri -jelly with PEITC intake dependent variable (outcome): adverse effects, health-related quality of life score, tumor response, progression-free survival, serum p53 and cytochrome C levels and functional status

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of squamous cell carcinoma in areas of lip, oral cavity, oropharynx and hypopharynx, who receive only palliative care or deny definitive treatment
2. Finished radiotherapy or/and chemotherapy for at least one month
3. Has at least one measurable target lesion
4. Baseline KPS ≥ 40% or ECOG 0-3
5. Blood tests are in acceptable ranges (neutrophils ≥ 1.5 x 109/L, platelets ≥ 100 x 109/L; Hb ≥ 9.0 g/dL), renal function (clearance creatinine using the CKD-EPI formula (Chronic Kidney Disease Epidemiology group) ≥50 mL/min) and hepatic function (SGOT , SGPT, serum bilirubin ≤ 1.5 of upper limits of normal
6. Able to take the intervention (through mouth or NG tube) without aspiration
7. Able to communicate and consent to the study

Exclusion Criteria:

1. Cannot come back for the follow-up visits
2. Receive or had received N-acetylcysteine during the intervention
3. Has systemic diseases that might interfere with the results
4. Chronic kidney disease that requires dialysis
5. Increased risk of aspiration pneumonia
6. Pregnancy or lactation
7. Untreated infectious diseases

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2014-08 (Actual); Primary Completion 2021-02 (Actual); Study Completion 2023-01 (Actual)

PRIMARY OUTCOMES:
Adverse events | 1 month and 3 months after receiving intervention
  Evaluation of adverse events by physical examination, blood tests, and interviewing the subjects
Changes in Health-related quality of life score compared to baseline | Baseline, 1 month and 3 months after receiving intervention
  Evaluation of Health-related quality of life by using questionnaire FACT-HN
Changes in Tumor response compared to baseline | Baseline, 1 month, 3 months after receiving intervention
  Evaluation of tumor response following RECIST criteria at 1 month and 3 months
Progression-free survival time | The time of the intervention until any signs or symptoms of progressive disease be recorded.
  The length of time during the intervention that the participant lives with stable disease

SECONDARY OUTCOMES:
Serum p53 level | 1 month and 3 months after receiving intervention
  Level of both wild type and mutant p53 in serum
Serum cytochrome C level | 1 month and 3 months after receiving intervention
  Level of cytochrome C in serum
Changes in Functional status | Baseline, 1 month and 3 months after receiving intervention
  Evaluation of functional status using KPS (Karnofsky Performance Score) score

CONTACTS AND LOCATIONS:
Overall Officials: Aroonwan Lam-ubol, DDS, PhD, Principal Investigator — Srinakharinwirot University
Locations (5):
- Thailand (5):
  - National cancer institute, Bangkok, Bangkok
  - Chonburi Cancer Hospital, Chon Buri, Changwat Chon Buri
  - Lopburi Cancer Hospital, Lopburi
  - Maharat Nakhon Ratchasima Hospital, Nakhon Ratchasima
  - Maha Vajiralongkorn Thanyaburi Hospital, Pathum Thani

IPD SHARING:
Plan to Share IPD: No